CLINICAL TRIAL: NCT04224103
Title: Nitric Oxide in Right Ventricular Dysfunction: Improvements in Clinical and Hemodynamic Parameters on Venoarterial Extracorporeal Membrane Oxygenation (VA-ECMO; NOVICE)
Brief Title: Nitric Oxide in Venoarterial Extracorporeal Membrane Oxygenation (VA ECMO)
Acronym: NOVICE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Filio Billia (Other)
Collaborators: Peter Munk Cardiac Center (Unknown); Heart and Stroke Foundation of Canada (Other); University of Toronto (Other)
Responsible Party: Sponsor-Investigator, Filio Billia, Director of Research, Peter Munk Cardiac Center, University of Toronto
Organization: University of Toronto (Other)
Other Study IDs: 15-8770
Record Dates: First submitted 2019-09-16; First posted 2020-01-13 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Extracorporeal Membrane Oxygenation; Nitric Oxide; Shock, Cardiogenic
Keywords: Venoarterial ECMO; VA-ECMO weaning; Inhaled nitric oxide; Right ventricle
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Inhaled nitric oxide
  Interventions: Drug: Inhaled nitric oxide

INTERVENTIONS:
Drug: Inhaled nitric oxide — Stage 1: Patients in whom VA ECMO is being initiated will be invited to participate. Hemodynamic, echocardiographic, and biochemical parameters will be measured immediately prior to iNO administration, and thirty minutes after initiation. After six hours, hemodynamic, echocardiographic, and biochemical parameters will be re-assessed after which iNO will be weaned. All parameters will be re-evaluated 30 minutes after iNO discontinuation.
  Stage 2: iNO will be re-initiated 30 minutes prior to the ECMO weaning trial. Hemodynamic, echocardiographic, and biochemical parameter will be recorded immediately prior to iNO administration and then at 30 minutes prior to the ECMO weaning trial. When ECMO weaning is unsuccessful, these parameters will be recorded immediately prior to re-initiation of full flow VA ECMO and 30 minutes thereafter. If successful, data will be collected after the wean and after iNO discontinuation.

SUMMARY:
This pilot study is designed to investigate the effect of inhaled nitric oxide on cardiac, pulmonary artery, and systemic hemodynamics at various time points during venoarterial extracorporeal membrane oxygenation (VA-ECMO) support. Patients who have been initiated on VA-ECMO will be invited to participate. Inhaled nitric oxide (iNO) will be used early after VA-ECMO cannulation (once consent is obtained). After baseline hemodynamic, biochemical, and echocardiographic parameters are assessed, iNO will be initiated and all parameters will be reassessed after 30 minutes and 6 hours. Inhaled nitric oxide will then be discontinued and all parameters repeated. At the time of VA-ECMO weaning (timing determined by clinical team), iNO will be reinitiated with repeat assessment of hemodynamic, biochemical, and echocardiographic parameters both prior to the wean and after the wean (whether successful or not).

DETAILED DESCRIPTION:
This is a proof of concept, pilot, phase II study using iNO in patients on VA-ECMO. Stage 1 will assess the participant's response to iNO early after cannulation. Stage 2 will assess the participant's response to iNO during the ECMO weaning process.

Stage 1 Patients in whom VA-ECMO is being initiated will be invited to participate. Hemodynamic, echocardiographic, and biochemical parameters will be measured immediately prior to iNO administration and repeated 30 minutes after iNO initiation. iNO will be continued for six hours to allow hemodynamic and oxygenation parameters to stabilize as per previous protocols in the literature. After six hours, hemodynamic, echocardiographic, and biochemical parameters will be re-assessed after which iNO will be discontinued. All parameters will be re-evaluated 30 minutes after iNO discontinuation.

Stage 2 A weaning trial will be performed at 1) the earliest signs of myocardial recovery or b) day 5. Myocardial recovery will be defined as: mean arterial pressure > 60 millimeters of mercury (mmHg) on no or minimal inotropic/vasopressor support, arterial pulse pressure > 10 mmHg, and minimal respiratory support (oxygen saturation > 88% on < 2 liters by nasal cannulae, or minimal ventilator setting if intubated). Inhaled nitric oxide will be re-initiated 30 minutes prior to the ECMO weaning trial. Adequacy of perfusion will be defined as a mixed venous oxygen saturation of > 70%. Hemodynamic, echocardiographic, and biochemical parameter will be recorded immediately prior to iNO administration and then at 30 minutes prior to the ECMO weaning trial. ECMO will be weaned as per the standard protocol at the University Health Network with re-assessment of all parameters after weaning is complete. When ECMO weaning is unsuccessful, these parameters will be recorded immediately prior to re-initiation of full flow VA-ECMO and 30 minutes thereafter. VA-ECMO weaning will be re-attempted at 24-48 hours at the discretion of the medical team.

ELIGIBILITY:
Inclusion Criteria:

* Age>18years
* History or evidence of left ventricular failure

Exclusion Criteria:

* ECMO cannulation site other than the femoral vein and artery
* Insufficient echocardiographic images to assess ventricular function
* Right ventricular assist device
* Uncorrected congenital heart disease
* Primary graft failure
* No cardiac output on bedside ECHO (LVEF<5%)
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of participants with decompensated heart failure in whom VA ECMO is being used as a bridge to recovery, cardiac transplantation, or durable mechanical circulatory support (MCS).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-08-08 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Participant recruitment | February 2020
  Recruitment of ten participants
Right Heart - Qualitative function, change from baseline | After 6 hours of inhaled nitric oxide
  Mild/moderate/severe dysfunction as determined by reading echocardiographer
Right Heart - Tricuspid annular plane systolic excursion (TAPSE), change from baseline | After 6 hours of inhaled nitric oxide
  Measured in milimeters
Right Heart - RV fractional area change, change from baseline | After 6 hours of inhaled nitric oxide
  Measured in percent
Right Heart - longitudinal myocardial velocity (S'), change from baseline | After 6 hours of inhaled nitric oxide
  Measured in meters per second

SECONDARY OUTCOMES:
Left Heart Function | After 6 hours of inhaled nitric oxide
  Left ventricular ejection fraction
Weaning success | Within 5 days of cannulation but may be repeated at 7 days if initially unsuccessful.
  Explore the effect of iNO on the rate of successful VA ECMO weaning.
Long-term RV function | Within three months of initial ECMO cannulation.
  Assess RV function after LVAD implantation or cardiac transplantation if these occur during the same hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Filio Billia, MD PhD, Principal Investigator — University of Toronto, Peter Munk Cardiac Centre
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No